CLINICAL TRIAL: NCT01980602
Title: A Randomised Controlled Trial to Analyse the Histological, Physiological and Haemorrheological Adaptations to Supervised Exercise Training in Claudicants
Brief Title: Effect of Exercise on Patients With Claudication Undergoing Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Hull (Other)
Responsible Party: Principal Investigator, Daniel Carradice, Academic Clinical Lecturer, University of Hull
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11/YH/0210
Record Dates: First submitted 2013-09-24; First posted 2013-11-11 (Estimated); Last update posted 2013-11-11 (Estimated); Status verified 2013-11

CONDITIONS: Intermittent Claudication; Peripheral Arterial Disease
Keywords: Intermittent claudication; endothelial function; cardiopulmonary testing; inflammation; muscle architecture
MeSH Terms: conditions — Intermittent Claudication; Peripheral Arterial Disease; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Supervised Exercise Program (Experimental)
  Interventions: Procedure: Supervised Exercise program

INTERVENTIONS:
Procedure: Supervised Exercise program

SUMMARY:
Title: How does exercise improve the calf muscle in patients with poor blood supply to their leg?

Purpose of the project: Patients with peripheral arterial disease have a poor blood supply to their lower leg. The reduced inflow prevents the leg from utilising nutrients and oxygen as easily as a healthy leg would. This causes pain when walking (intermittent claudication), which often occurs after a reproducible distance e.g. every 50 yards. These patients have a reduction in their quality of life as they feel embarrassed in social situations e.g. walking around town requires multiple breaks, so they tend to avoid this and isolate themselves more.

One treatment for claudication is exercising until the pain comes on; which most are reluctant to do. Walking up to three times a week for an hour, can double most people's walking distances, but doesn't always. The reason why some improve with exercise and others do not remains unknown.

This project will be the first randomised controlled trial of exercise in claudicants that focuses on the adaptations that occur in the muscle at a cellular level. We wish to compare muscle cells from a group that have exercised and group that have not. We will focus on the change in muscle cell size and function at present, and later progress to why and how this happens.

Methods: We will take measurements at the start of the study (baseline), after 6 weeks and then 3, 6 and 12 months. These measurements will be of a patient's fitness, actual walking distances and blood samples. At the time of surgery, muscle from the calf will be taken from the affected leg. This will be processed at the University's biomedical science department to look at the different types of muscle fibre and how efficiently they are working.

ELIGIBILITY:
Inclusion Criteria:

* Community dwelling older adults aged 45 and over
* Diagnosis of intermittent claudication - ABPI < 0.9 with symptoms in keeping with intermittent claudication
* Undergoing surgery for claudication
* Ability to walk without assistance
* Healthy control patients who are undergoing varicose vein surgery

Exclusion Criteria:

* Participants who are unable to provide informed consent
* Severe of acute cardiovascular, musculoskeletal or pulmonary illness
* Critical limb ischaemia
* Active treatment for cancer
* Rheumatoid arthritis or any patient receiving steroids or disease modifying Antirheumatic drugs (DMARDS)
* Failure to complete a CPET

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2011-03; Primary Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Measurement of cardiovascular ability as recorded by their anaerobic threshold and peak VO2 after 6 weeks of exercise training or standard care | 6 weeks
  Patients will undergo cardiopulmonary exercise testing to assess whether a 6 week exercise programme improves the cardiovascular fitness

SECONDARY OUTCOMES:
Measure the changes in muscle fibre type with exercise training or standard care | Baseline, 6 weeks, 3 months, 6 months, and 12 months
  Histological analysis to measure the percentage of different types of muscle fibres, and how these are affected by 6 weeks of exercise compared to standard treatment.
Measurement of endothelial function after a period or exercise therapy or standard care | Baseline, 6 weeks, 3 months, 6 months, and 12 months
  To identify if 6 weeks of exercise improves the endothelial function.
Measurement of inflammatory markers with exercise treatment or standard care | Baseline, 6 weeks, 3 months, 6 months, and 12 months
  To identify whether 6 weeks of exercise therapy improves inflammatory markers

CONTACTS AND LOCATIONS:
Overall Officials: Romesh Sarvanandan, MBBS MRCS, Principal Investigator — Hull York Medical School/ University of Hull/ Hull and East Yorkshire NHS Trust
Locations (1):
- Hull Royal Infirmary, Hull, United Kingdom